CLINICAL TRIAL: NCT06934707
Title: Meal Frequency, Glycemic Control and Variability in Individuals With Type 1 Diabetes: a Randomized Crossover Clinical Trial
Brief Title: Meal Frequency and Glycemic Control in Individuals With Type 1 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0583; 2022-0583 (Other Grant/Funding Number: FIPE/HCPA)
Record Dates: First submitted 2025-03-20; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes (T1D); Nutrition Therapy; Glycemic Control for Diabetes Mellitus
Keywords: type 1 Diabetes; glycemic control; diet; meal frequency
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Each intervention phase will span 3 weeks, followed by a 4-week washout phase.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The participants and the care providers will not be blinded. People involved in assessing outcomes and with data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 meals a day (Experimental): Diet for maintaining body weight with three meals per day
  Interventions: Behavioral: Three meals a day
- 6 meals a day (Active Comparator): Diet for maintaining body weight with six meals a day
  Interventions: Behavioral: Six meals a day

INTERVENTIONS:
Behavioral: Three meals a day — This group will follow a dietary prescription consisting of three meals per day. The total energy value will be distributed in accordance with the macronutrient recommendations for type 1 diabetes (T1D), as follows: 45% of energy from total carbohydrates, prioritizing those with a low glycemic index; up to 30% from total fats, with unsaturated fats being the primary source; and 25% of energy from proteins. Caloric distribution will be divided into 30% for breakfast, 40% for lunch, and 30% for dinner, with 14 g of fiber per 1000 kcal distributed across the three meals. Furthermore, the gram amounts of the macronutrient in each meal will be apportioned such that 15-20% of the total carbohydrate intake, 7-10% of the total protein intake, and 10% of the total fat intake.Participants will also be instructed to maintain their habitual physical activity level.
  Arms: 3 meals a day
Behavioral: Six meals a day — This group will follow a dietary prescription consisting of six meals per day. The total energy value will be distributed in accordance with the macronutrient recommendations for type 1 diabetes (T1D), as follows: 45% of energy from total carbohydrates, prioritizing those with a low glycemic index; up to 30% from total fats, with unsaturated fats being the primary source; and 25% of energy from proteins. Caloric distribution will be divided into 20% for breakfast, 10% morning snack, 30% for lunch, 10% afternoon snack, 25% for dinner and 5% bedtime snack, with 14 g of fiber per 1000 kcal distributed across the three meals. Furthermore, the gram amounts of the macronutrient in each meal will be apportioned such that 5-10% of the total carbohydrate intake, 2-7% of the total protein intake, and 2-8% of the total fat intake.Participants will also be instructed to maintain their habitual physical activity level.
  Arms: 6 meals a day

SUMMARY:
The goal of this clinical trial is to examine the effect of 3 versus 6 daily meals of isocaloric diets on glycemic control and variability in individuals with type 1 diabetes. Participants will be randomized in a crossover clinical trial and will receive two different types of isocaloric diet interventions, in 3 meals/day (calorie distribution: 30% at breakfast, 40% at lunch and 30% at dinner) or 6 meals/day (calorie distribution: 20% at breakfast, 10% at morning snack, 30% at lunch, 10% at afternoon snack, 25% at dinner and 5% at evening snack), for three weeks, with a 4-week washout period between diets.

DETAILED DESCRIPTION:
This is a single center, randomized, open-label, non-inferiority and crossover clinical trial. Subjects with type 1 diabetes (T1D) and will be recruited through advertisement on the web page of Hospital de Clínicas de Porto Alegre (HCPA), type 1 diabetes outpatient clinic of HCPA, local newspaper, television and social media, or referred by a doctor or nutritionist, from external to HCPA services. After screening and selection according to inclusion criteria, participants will undergo a clinical, laboratory and nutritional evaluation following a standard assessment protocol. After all baseline assessments, they will be randomly allocated to one of the following interventions for 3 weeks and after a washout period, they will be in the other intervention. While glycemic control (A1c and Glycated albumin) and variability (6 points daily capillary blood glucose tests) are assessed during the baseline period, the first week of each intervention, and the last week of washout and continuous interstitial glucose measurements that are performed in the last 14 days of each intervention. Blinding is maintained outcome assesment.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (18 to 60 years old) with a medical diagnosis of type 1 diabetes mellitus

  * Individuals who perform carbohydrate counting
  * Individuals diagnosed > 12 months ago
  * Perform daily glycemic control using a blood glucose monitor or use of a glucose sensor
  * Have the ability to understand and be able to adhere to the proposed interventions.
  * Complete a detailed 3-day food record for one week prior to the intervention and record episodes of hypoglycemia (<70 mg/dL) and hyperglycemia (>180 mg/dL)
  * Able and willing to provide written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

* Individuals with glycated hemoglobin ≥ 11%
* Individuals who are using NPH insulin
* Retinopathy with vision deficit that limits the activities proposed in the disciplines.
* Individuals with gastrointestinal disease such as celiac disease, Crohn's disease and Irritable Bowel Syndrome (IBS)
* History of bariatric surgery
* That you are following a carbohydrate, protein and/or fat restriction diet
* Individuals with BMI ≥ 40kg/m2
* Chronic kidney disease with estimated glomerular filtration <30mL/min per 1.73 m2.
* Liver failure or chronic viral hepatitis
* Active or progressive neurodegenerative disease
* Use of medications that affect glucose metabolism (corticosteroids and immunosuppressants) or cause weight loss. ● Treatment with weight-reducing agents (e.g., orlistat, sibutramine, topiramate, liraglutide) in the last 12 weeks prior to screening.
* Treatment with thyroid hormone that has not been maintained at a stable dose in the last 12 weeks prior to screening.
* History of active substance abuse (including alcohol) in the last year.
* Serious psychiatric illness: Mood disorders, anxiety disorders, severe psychotic disorders, and personality disorders that are revealed or identified in the clinical evaluation, listed or reported in the medical record, and that have no clinical findings.
* Predisposition to or diagnosis of eating disorders.
* Women who are pregnant, intending to become pregnant during the study period, or who are breastfeeding.
* Hyperglycemia characterized by acute symptoms: polyuria, polydipsia, and/or weight loss in the last 3 months. ● Metabolic and acute complications of diabetes such as ketoacidosis or hyperosmolar coma.
* Night workers who work after 10 pm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-12-29 (Estimated); Study Completion 2027-12-29 (Estimated)

PRIMARY OUTCOMES:
Change in glycemic control | Baseline, 5, 6, 12 and 13 weeks
  Differences Between Groups in Glycemic Control and Variability Using HbA1c and Freestyle Libre Continuous Glucose Monitoring (CGM)

SECONDARY OUTCOMES:
Change in Glycated Hemoglobin | Baseline, 3, 6, 10 and 13 weeks
  Difference between groups in glycated hemoglobin
Glycemic Variability | 5 and 12 weeks
  For continuous glucose monitoring and assessment of glycemic variability, the FreeStyle Libre, ABBOTT® device will be used. FreeStyle Libre consists of a continuous glucose monitoring (SMCG) system. Glycemic variability will be assessed using time on target parameters of values between 70 and 180 mg/dL, values between 70 and 140mg/dL, time in hypoglycemia and time above target and coefficient of variability as measures of glycemic variability
Changes in body composition | Baseline, 3, 6, 10 and 13 weeks
  Weight, fat-free mass and fat mass will be assessed by Bioelectrical Impedance (body composition analyzer tetrapolar InBody 370S, BiospaceCo. Ltd, Seoul, South Korea). Anthropometric measures include brachial, neck, waist, hip and calf circumferences, with participants wearing light clothing and barefoot.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Gerchman, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No